CLINICAL TRIAL: NCT04411108
Title: Validation of Motion Coaching Technology for Physical Therapy in Treating Patients With Chronic, Nonspecific Low Back Pain. A Pilot Project.
Brief Title: Motion Coaching Technology for Physical Therapy in Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaia Health Software (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KaiaMC001
Record Dates: First submitted 2020-05-14; First posted 2020-06-02 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Instruction by PT and written handout (Active Comparator)
  Interventions: Other: Physiotherapist Exercise Instructions and written handouts
- Exercise Instruction by Motion Coach Technology (Experimental)
  Interventions: Other: Kaia Back Pain App

INTERVENTIONS:
Other: Kaia Back Pain App — The Kaia Back Pain App provides instructions on exercise execution to participants for one week
  Arms: Exercise Instruction by Motion Coach Technology
Other: Physiotherapist Exercise Instructions and written handouts — Participants will be instructed by physiotherapists in exercise execution and receive handouts and exercise for one week
  Arms: Exercise Instruction by PT and written handout

SUMMARY:
In this study, we will compare exercise execution between two groups of patients: (1) individuals who undergo instruction session by a PT and then perform exercises with a written handout at home and (2) individuals who use the mHealth motion coach at home. Participants will perform the same 4 exercises. Both groups will be instructed to exercise at home, supported either by the handouts or the Motion Coach technology and then return after 1 week for assessment.

For the assessment, standardized videos will be used to capture pose during exercise execution. Group 1 will perform the exercises with the written handout; group 2 will perform the exercises with the motion coach. Rating will be performed by a panel of PT professionals on the overall assessment of each exercises and on the three segments mentioned below that are exercise specific. The first group with PT instruction and written handout portion will be compared to the second group with the motion coach.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 - 65
* English speaking
* Absence of neurologic deficits as assessed by the clinician, with 5/5 strength in all muscle groups in the lower extremities and no sensory deficits in the lower extremities
* Pain located in the low back or posterior pelvic region
* Self-reported mean pain score >4 in the past 1 week as assessed by VAS pain score from 0-10
* Pain duration >1 month to 5 years
* Ambulatory w/out assist prior to enrollment

Exclusion Criteria:

* Red flag signs including fevers, unexplained weight loss, personal history of cancer, tuberculosis exposure, history of spinal infection, history of thoracolumbar spine fracture in the past year as assessed by the clinician.
* Use of assistive ambulatory device
* Pregnancy
* Formal physical therapy within the past 6 months
* Neurologic symptoms including weakness or sensory changes in the bilateral lower extremities as assessed by the clinician.
* Pain radiating below the posterior pelvic region into either lower extremity
* Unwilling or unable to commit to study procedures
* Physically incapable of completing PT exercises safely as determined by clinician

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Scoring of each individual exercise rated by a panel of physiotherapists | 7 days
  A panel of 5 physiotherapists each rates every repetition recorded as acceptable or not. If greater than 90% are rated as acceptable, the exercise will be assessed as acceptable.

SECONDARY OUTCOMES:
Rating of exercise execution concerning specific body regions by physiotherapists | 7 days
  For predefined segments for every exercise, a panel of physiotherapists scores execution quality on a scale of 0-3

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedic Surgery, Division of Spine Surgery, Washington University in St. Louis, MO, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No